CLINICAL TRIAL: NCT04358497
Title: Endovascular Versus Medical Treatment for the Pelvic Congestion Syndrome
Acronym: ENDPCS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clínicas Dr. Manuel Quintela (Other)
Collaborators: University of the Republic, Uruguay (Other); Centro Cardiovascular Universitario (Unknown); Centro Hospitalario Pereyra Rossell (Unknown)
Responsible Party: Principal Investigator, Eduardo Sebastian Sarutte Rosello, MD VS MSc, Vascular Surgery Asistant Professor, Hospital de Clínicas Dr. Manuel Quintela
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TR001
Record Dates: First submitted 2020-01-17; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Pelvic Congestive Syndrome; Pelvic Varices; Venous Disease
Keywords: pelvic congestion syndrome; sclerosis; coil embolization
MeSH Terms: conditions — Sclerosis | interventions — Diosmin; Hesperidin; Ibuprofen; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Intervention Model Description: Blind randomized clinical trial designed to compare the efficacy and safety of endovascular treatment of Pelvic congestion syndrome.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Phlebography will be performed to both groups. On the experimental group, the treatment of the pelvic congestion will be performed, while the procedure will be stopped on the control group. Neither the patient or the reference gynecologist will be informed if the treatment took place.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Interventional treatment plus best chronic medical treatment (Experimental): Sandwich embolization ( 2% polidocanol + Coils) Diosmin hisperidin 1g twice a day for 6 months Ibuprofen 500mg 3 times a day for 6 months
  Interventions: Device: Medtronic® Concerto® detachable coil system; Procedure: sclerosis; Drug: Diosmin / Hesperidin; Drug: Ibuprofen 400 mg
- Best chronic medical treatment alone (Active Comparator): Diosmin hisperidin 1g twice a day for 6 months Ibuprofen 500mg 3 times a day for 6 months
  Interventions: Drug: Diosmin / Hesperidin; Drug: Ibuprofen 400 mg

INTERVENTIONS:
Device: Medtronic® Concerto® detachable coil system — coil embolization of the reflux pathways
  Other Names: concerto detachable coil system
  Arms: Interventional treatment plus best chronic medical treatment
Procedure: sclerosis — Pelvic varices sclerosis with polidocanol foam
  Other Names: Foam sclerosis with polidocanol 2%
  Arms: Interventional treatment plus best chronic medical treatment
Drug: Diosmin / Hesperidin — Best chronic medial treatment
  Other Names: daflon
Drug: Ibuprofen 400 mg — NSAID treatment
  Other Names: Nsaid

SUMMARY:
Compare the efficacy and safety of endovascular treatment with sandwich technique (controlled release coils and 2% polidocanol foam) associated with diosmin-hisperidine and ibuprofen medical treatment and only the best chronic medical treatment available diosmin-hisperidine and ibuprofen for 3 months, in women of active gynecological age carrying pelvic congestion syndrome in public assistance in Montevideo, Uruguay.

DETAILED DESCRIPTION:
Pelvic congestion syndrome (PCS) is a recognized and frequent cause of Chronic Pelvic Pain (10% to 30%). It is defined as the presence of chronic symptoms, which may include pelvic pain, perineal heaviness, urinary urgency and postcoital pain, caused by reflux and / or obstruction of the gonadic and / or pelvic veins, and that may be associated with vulvar, perineal and lower limbs varicose veins.

There is no standard approach to managing PCS. According to expert recommendations, therapies should be individualized according to the patient's symptoms and needs.

Medical treatment options include progestagens, danazol, combined oral hormonal contraceptives, phlebotonics such as hisperidine-added diosmin, non-steroidal anti-inflammatory drugs and gonadotropin-releasing hormone (GnRH) agonists

Currently, the only accepted chronic medical treatment is the association of non-steroidal and phlebotonic anti-inflammatories, but they have shown a poor symptomatic benefit in reducing pain.

Surgical treatment has evolved over time mainly in the hands of laparoscopic techniques, currently the endovascular option is the most widely accepted for presenting excellent long-term results with abolition of pain in up to 90% at 2 years.

HYPOTHESIS

Endovascular treatment of pelvic congestion syndrome is better in terms of pain control and quality of life compared to drug treatment.

General objective

Compare the efficacy and safety of endovascular treatment with sandwich technique (controlled release coils and 2% polidocanol foam) associated with diosmin-hisperidine and ibuprofen medical treatment and only the best chronic medical treatment available diosmin-hisperidine and ibuprofen for 3 months, in women of active gynecological age carrying pelvic congestion syndrome in public assistance in Montevideo, Uruguay.

Specific objectives

• Compare pain in patients undergoing endovascular treatment with the best

medical treatment.

* Evaluate the persistence of pelvic varices in patients undergoing endovascular treatment of SCP.
* Compare the Female Sexual Satisfaction Index in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Active gynecological age
* Chronic pelvic pain diagnosed by gynecologist of at least 6 months of evolution.
* Transvaginal duplex ultrasound: presence of periuterine varicose veins defined by veins larger than 5mm in diameter with reflux greater than 0.5 seconds on Valsava maneuvers.

Exclusion Criteria:

* Presence of other causes of chronic pelvic pain: endometriosis, pelvic inflammatory disease, postoperative adhesions, uterine myoma, adenomyosis, ovarian tumors, polycystic ovary.
* Fibromyalgia
* BMI greater than 35
* Chronic kidney disease
* thrombophilia
* Alterationof coagulation.
* Allergy to iodinated contrast medium.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale (VAS) | 30 days
  Pain assessment 1-10 from no pain to severe
visual analogue scale (VAS) | 3 months
  Pain assessment 1-10 from no pain to severe
Lattinen index | 30 days
  chronic pain assessment 2-22 from low to high
Lattinen index | 3 months
  chronic pain assessment 2-22 from low to high
McGill Pain Questionnaire | 30 days
  subjective pain experience assessment
McGill Pain Questionnaire | 3 months
  subjective pain experience assessment

SECONDARY OUTCOMES:
Female sexual function index | 30 days
  questionnaire that assesses different domains of sexual function. 0-48 from no sexual distress to high level of sexual distress
Female sexual function index | 3 months
  questionnaire that assesses different domains of sexual function. . 0-48 from no sexual distress to high level of sexual distress
varicose and reflux persistance by transabdominal duplex scan | 30 days
  transabdominal duplex scan: varicose permeability, prescience of gonadic or iliac reflux
varicose and reflux persistance by transabdominal duplex scan | 3 months
  transabdominal duplex scan: varicose permeability, prescience of gonadic or iliac reflux
varicose and reflux persistance by transvaginal duplex scan | 3 months
  transabdominal duplex scan: varicose permeability, prescience of gonadic or iliac reflux
varicose persistance assesment by tomography | 3 months
  angiotomography: Varicose and conadic Patency

OTHER OUTCOMES:
Deep venous thrombosis by duplex ultrasound | 30 days
  Deep venous thrombosis of the iliac or femoral axis will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Sarutte, VS, Principal Investigator — Centro Cardiovascular Universitario

IPD SHARING:
Plan to Share IPD: Yes
De-identified data base for all variables will be available for researchers
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From April 2022 to april 2024
Access Criteria: Data will be shared on request, after signing a discretion agreement.